CLINICAL TRIAL: NCT06968208
Title: Randomized Controlled Trial of Puerarin for Obesity Treatment
Brief Title: The Efficacy and Safety of Puerarin in Obesity Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ruijin2025-177
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Diseases; Obesity/Therapy
Keywords: Puerarin; Intestinal Lipid Absorption; Dorsal Motor Nucleus of Vagus (DMV)
MeSH Terms: conditions — Metabolic Diseases; Obesity | interventions — puerarin

STUDY DESIGN:
Intervention Model Description: This study utilizes a randomized, double-blind, placebo-controlled, parallel-group design. Participants will be allocated 1:1 to either the intervention group receiving daily oral puerarin (75 mg/day, dissolved in 100 mL of 0.9% sodium chloride solution) or the control group receiving identically matched blank 100 mL of 0.9% sodium chloride solution for 6 consecutive months. Randomization will be stratified by baseline body mass index (BMI) and performed via a centralized computer-generated sequence with allocation concealment. Both participants and investigators will remain blinded to treatment assignment throughout the trial. Primary efficacy endpoints (body weight reduction, waist circumference, and lipid profile improvement) and safety outcomes (adverse events, hematological/biochemical parameters) will be assessed at baseline, 1, 3, and 6 months post-randomization. The study adheres to CONSORT guidelines for clinical trial reporting.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puerarin Group (Experimental): 1. Diet Stabilization (Days 0-3): Standardized high-fat isocaloric diet (25% carbs, 58% fat, 17% protein) to normalize baseline metabolic status.
  2. Intervention Period (6 months): Participants will receive oral administration of 75 mg puerarin dissolved in 0.9% sodium chloride solution, taken 30 minutes before lunch
  Interventions: Drug: Puerarin
- Placebo Group (Placebo Comparator): 1. Diet Stabilization (Days 0-3): Standardized high-fat isocaloric diet (25% carbs, 58% fat, 17% protein) to normalize baseline metabolic status.
  2. Intervention Period (6 months): Participants will receive oral administration of one matching blank 0.9% sodium chloride solution, taken 30 minutes before lunch. Blank injections are identical in appearance, taste, and packaging to the active puerarin injections but contain no active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Puerarin — 75 mg of puerarin injection, dissolved in 0.9% sodium chloride solution. The puerarin injection is manufactured under Good Manufacturing Practice (GMP) conditions by [Harbin Medisan Pharmaceutical Co., Ltd.], with identical appearance, size, and packaging to the blank 0.9% sodium chloride solution to ensure blinding. Stability testing confirms integrity under standard storage conditions (25°C, 60% RH).
  Arms: Puerarin Group
Drug: Placebo — 0.9% sodium chloride solution formulated to match the appearance, size, and taste of the active puerarin solution, with no other active pharmaceutical ingredients. 0.9% sodium chloride solution is manufactured under identical Good Manufacturing Practiceconditions by [Shijiazhuang No.4 Pharmaceutical Co., Ltd.] and changed to the same batch processes and packaging as the intervention group. Stability testing confirms equivalent integrity under standard storage conditions (25°C, 60% RH). Blinding is ensured through indistinguishable outer packing characteristics and labeling.
  Arms: Placebo Group

SUMMARY:
This randomized controlled trial aims to evaluate the therapeutic efficacy of puerarin intervention in weight management and metabolic regulation among obese populations. The study will systematically address two primary endpoints: 1) The capacity of puerarin to induce clinically significant body weight reduction in individuals with BMI ≥30 kg/m²; 2) Its modulatory effects on postprandial lipid metabolism as measured by serum lipids and quantitative fecal lipid excretion analysis. Secondary outcomes focus on puerarin's pleiotropic effects, including continuous glucose monitoring-derived glycemic parameters and indirect calorimetry-assessed resting metabolic rate. Secondary exploratory objectives include investigating puerarin's potential mechanisms of action through continuous glucose monitoring and indirect calorimetry measurements to assess glycemic variability and resting energy expenditure, respectively. Participants will be randomized into two parallel groups: the intervention group receiving daily oral puerarin injection (75 mg/day, dissolved in 100 mL of 0.9% sodium chloride solution) and the control group receiving matched blank 100 mL of 0.9% sodium chloride solution, both administered double-blind for 6 consecutive months. Primary efficacy endpoints (body weight, waist circumference, lipid profile) and safety monitoring (adverse events, hematological/ biochemical parameters) will be assessed at baseline, 1, 3, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years (inclusive), any gender.
2. Obesity (BMI ≥30.0 kg/m²).
3. With or without obesity-related metabolic comorbidities (e.g., type 2 diabetes, hypertension, dyslipidemia, hyperuricemia).
4. No prior use of weight-control, glucose-lowering, or lipid-modifying medications.
5. Stable weight (<3% fluctuation) and lifestyle for ≥1 month prior to screening.
6. Fully informed of trial objectives, procedures, risks, and benefits; voluntarily signed informed consent form.

Exclusion Criteria:

1. Secondary causes of obesity (e.g., monogenic obesity, Cushing's syndrome, drug-induced obesity).
2. History of common nutrient allergies (e.g., gluten, milk, eggs, plant-derived proteins).
3. Use of weight-control medications (e.g., metformin, GLP-1 receptor agonists, orlistat), corticosteroids (oral/IV/IM/non-oral systemic/intra-articular), or metabolic-interfering drugs/supplements within 3 months prior to screening or during the trial.
4. Use of traditional Chinese medicines or herbal products for weight management within 3 months prior to screening or during the trial.
5. History of psychiatric disorders, epilepsy, antidepressant use, or ongoing antiepileptic therapy.
6. Pregnancy, lactation, or plans for pregnancy within 6 months post-trial.
7. Active infectious diseases (e.g., HBV, HCV, tuberculosis, syphilis, HIV).
8. Severe infections, severe anemia (Hb <8 g/dL), or neutropenia (ANC <1.5×10⁹/L).
9. Gastrointestinal surgery within 1 year (excluding appendectomy/hernia repair) or major non-GI surgery within 6 months.
10. Active substance/alcohol abuse.
11. Known hypersensitivity to trial drug components or history of severe drug allergies.
12. Severe cardiac disorders (e.g., congenital/rheumatic heart disease, cardiomyopathy [NYHA ≥III], coronary stenting).
13. Hyperthyroidism or hypothyroidism.
14. History of malignancies (treated/untreated), regardless of recurrence status.
15. Hepatic/renal dysfunction: ALT/AST ≥2.5×ULN, serum creatinine >ULN, or eGFR <60 mL/min/1.73m² (MDRD formula).
16. Gastrointestinal disorders affecting absorption (e.g., IBD, active ulcers, severe diarrhea/constipation).
17. Participation in other clinical trials within 3 months prior to screening.
18. Any condition deemed unsuitable by investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.
  Body weight will be measured to the nearest 0.1 kg using a calibrated digital scale under standardized conditions: participants in lightweight clothing (hospital gown), barefoot, and after an overnight fast (≥8 hours).
Body Fat Percentage | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.
  Body fat percentage will be quantified via bioelectrical impedance analysis (BIA, InBody 770®).
Serum Lipid Profile (Total Cholesterol [TC], Triglycerides [TG]) | Measurements will be performed at each timepoint (baseline, 1, 3, and 6 months post-intervention) and twice a day
  Total Cholesterol (TC): Measured via cholesterol oxidase-peroxidase method, traceable to CDC reference standards. Triglycerides (TG): Quantified using glycerol-3-phosphate oxidase method with correction for free glycerol. The blood samples will be collected before and 2 hours after meals.
Fecal Lipids | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.

SECONDARY OUTCOMES:
Blood Glucose | Measurements will be performed at each timepoint (baseline, 1, 3, and 6 months post-intervention) and twice a day
  The blood samples will be collected after overnight fasting and 2 hours after meals.
Basal Metabolic Rate | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.
  Basal metabolic rate will be measured via indirect calorimetry using a validated metabolic cart under strictly standardized conditions: participants in a fasting state (≥12 hours overnight), resting supine in a thermoneutral environment (22-24°C), with 30 minutes of pre-measurement rest and avoidance of caffeine or vigorous activity for 24 hours prior.
Gut Hormones | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.
  Like ghrelin, cholecystokinin (CCK), Glucagon-like peptide-1 (GLP-1), Peptide YY (PYY)
Insulin level | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.
  The blood samples will be collected after overnight fasting(>8 hors).
Gut Microbiome Metagenomics | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention).
C-Peptide | Measurements will be performed in quadruplicate at each timepoint (baseline, 1, 3, and 6 months post-intervention), with the mean value recorded.
  The blood samples will be collected after overnight fasting(>8 hors).

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No